CLINICAL TRIAL: NCT04089371
Title: A Post-Market Clinical Evaluation of the ReUnion Reversible Fracture (RFX) System
Status: Terminated | Type: Observational
Why Stopped: Sponsor Terminated
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Other Study IDs: ReUnion RFX Study
Record Dates: First submitted 2019-07-11; First posted 2019-09-13 (Actual); Results first posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Arthroplasty; Hemiarthroplasty; Shoulder Pain
Keywords: Arthroplasty; Hemiarthroplasty; Shoulder; Replacement
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Arm A Total Shoulder Arthroplasty / Hemiarthroplasty: Total Shoulder Arthroplasty (TSA) Humeral & Glenoid components as a Hemiarthroplasty or Total Shoulder Replacement.
  Interventions: Device: ReUnion Total Shoulder Arthroplasty (TSA)
- Arm B Reverse Shoulder Arthroplasty: Reverse Shoulder Arthroplasty (RSA) Humeral & Glenoid Components as a primary, fracture or revision total shoulder replacement
  Interventions: Device: ReUnion Reverse Shoulder Arthroplasty (RSA)

INTERVENTIONS:
Device: ReUnion Total Shoulder Arthroplasty (TSA) — The ReUnion RFX System includes a Reversible Fracture Stem (RFX Stem) that can utilize either the ReUnion Total Shoulder Arthroplasty (TSA) or ReUnion Reverse Shoulder Arthroplasty (RSA) humeral and glenoid components and is indicated for use as a hemi, total or reverse shoulder replacement. The ReUnion RFX stem is intended for cemented use only.
  Groups: Arm A Total Shoulder Arthroplasty / Hemiarthroplasty
Device: ReUnion Reverse Shoulder Arthroplasty (RSA) — The ReUnion RFX System includes a Reversible Fracture Stem (RFX Stem) that can utilize either the ReUnion Total Shoulder Arthroplasty (TSA) or ReUnion Reverse Shoulder Arthroplasty (RSA) humeral and glenoid components and is indicated for use as a hemi, total or reverse shoulder replacement. The ReUnion RFX stem is intended for cemented use only.
  Groups: Arm B Reverse Shoulder Arthroplasty

SUMMARY:
This investigation is a prospective, multi-center clinical investigation. It is anticipated that a total of one hundred (100) subjects will be enrolled at approximately 5-10 sites. The clinical investigation has been designed to follow the surgeon's standard of care for joint arthroplasty patients, which entails clinical evaluation on a regular ongoing basis, or as needed should the patient become symptomatic in the treated joint.

DETAILED DESCRIPTION:
The objective of this clinical investigation is to demonstrate the safety and efficacy/performance of the ReUnion RFX System. Efficacy/performance of the procedure will be measured by the American Shoulder and Elbow Surgeons (ASES) Shoulder Score. Safety of the ReUnion RFX System will be demonstrated through reporting of device-related intraoperative and postoperative Adverse Events (AEs). Enrolled subjects will be assessed at Pre-Operative, Operative/Discharge, and at 6 Weeks, 6 Months, 12 Months, 24 Months and annually thereafter up to 10 years following the index procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing to sign the informed consent.
* Subject is willing and able to comply with postoperative scheduled clinical evaluations.
* Subject is male or non-pregnant female and 18 years or older at the time of surgery.
* When used with ReUnion Total Shoulder Arthroplasty (TSA)Humeral & Glenoid components as a Hemiarthroplasty or Total Shoulder Replacement, subject has one or more of the following:

  * Aseptic necrosis of humeral head;
  * Painful, disabling joint disease of the shoulder resulting from degenerative arthritis, rheumatoid arthritis or post-traumatic arthritis;
  * Proximal humeral fracture and/or dislocation;
  * Clinical management problems where arthrodesis or alternative reconstructive techniques are less likely to achieve satisfactory results;
  * Previous unsuccessful total shoulder replacement, resurfacing or other procedure
* When used with ReUnion RSA Humeral & Glenoid Components as a primary, fracture or revision total shoulder replacement, subject's joint has gross rotator cuff deficiency, a functional deltoid muscle and is anatomically and structurally suited to receive the implant, and subject has one or more of the following:

  * Painful, disabling joint disease of the shoulder resulting from degenerative arthritis or rheumatoid arthritis;
  * Proximal humeral fracture
  * Previously failed shoulder joint replacement

Exclusion Criteria:

* Subject has an active or suspected latent infection in or about the shoulder joint.
* Subject has mental or neuromuscular disorder which would create an unacceptable risk of prosthesis instability, prosthesis fixation failure or complications in postoperative care.
* Subject has bone stock compromised by disease, infection or prior implantation which cannot provide adequate support and/or fixation to the prosthesis.
* Subject has anticipated activities which would impose high stresses on the prosthesis and its fixation.
* Subject is obese such that he/she produces a load on the prosthesis which can lead to failure of fixation of the device or to failure of the device itself.
* Subject has severe concomitant disease(s)which may significantly affect the clinical outcome.
* For Total Shoulder Arthroplasty and Hemiarthroplasty: Subject has absent, irreparable or non-functioning rotator cuff and other essential muscles

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects participating in this clinical investigation will be recruited from the investigator's standard patient population, where patients will be evaluated for clinical investigation participation based on the eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Gibson, Study Director — Stryker Trauma
Locations (3):
- United States (3):
  - Great Plains Orthopaedics, Peoria, Illinois
  - Steadman Hawkins, Greenville, South Carolina
  - Tennessee Orthopaedic Alliance, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A Total Shoulder Arthroplasty / Hemiarthroplasty | Arm B Reverse Shoulder Arthroplasty
Started | 0 | 10
Completed | 0 | 0
Not Completed | 0 | 10
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Study terminated early | 0 | 9

BASELINE CHARACTERISTICS:
Population: No cases were enrolled under Arm A
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A Total Shoulder Arthroplasty / Hemiarthroplasty | Arm B Reverse Shoulder Arthroplasty | Total
Number analyzed (Participants) | 0 | 10 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 70.80 (7.64) | 70.80 (7.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 9 | 9
  Male |  | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Caucasian |  | 10 | 10
  Ethnicity: N/A |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 10 | 10
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] |  | 30.62 (6.67) | 30.62 (6.67)

OUTCOME MEASURES:

1. Primary Outcome: 24-month Mean ASES Shoulder Score: Arm B (Reverse Shoulder Arthroplasty)
Description: This is a mixed outcome reporting measure, applicable for use in patients with shoulder pathology regardless of diagnosis and consists of a pain visual analog scale (VAS) and 10 functional questions. The primary endpoint of the clinical investigation is to demonstrate non-inferiority of the device to the selected literature controls, as measured by the ASES Shoulder Score at 24 Months post-operative. Scores range from 0 to 100 with a score of 0 indicating a worse shoulder condition and 100 indicating a better shoulder condition.
Time Frame: 24 months
Population: No Subjects were enrolled in Arm A. *Limited Sample Size for Arm B at 24mths, only 2 out of 10 subjects with available data for Arm B.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm B Reverse Shoulder Arthroplasty
Number analyzed (Participants) | 2
score on a scale | 86.50 (4.95)

2. Primary Outcome: 12-month Mean ASES Shoulder Score: Arm B (Reverse Shoulder Arthroplasty)
Description: as for outcome 1
Time Frame: *12 months (reporting 12mth as more data available)
Population: No Subjects were enrolled in Arm A. *Limited Sample Size for Arm B at 12mths, only 4 out of 10 subjects with available data for Arm B.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm B Reverse Shoulder Arthroplasty
Number analyzed (Participants) | 4
score on a scale | 65.25 (20.82)

3. Secondary Outcome: Device-related Adverse Events
Description: Incidence of intraoperative and post-operative adverse events related to the device will be collected and reported. Time to earliest device-related incident will be analyzed.
Time Frame: 24 mths
Population: No adverse events were reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm B Reverse Shoulder Arthroplasty
Number analyzed (Participants) | 10
Participants | 0

4. Secondary Outcome: Implant Survivorship
Description: Time to mortality or last available assessment will be measured and reported.
Time Frame: 10 years
Population: Due to early study termination, the planned implant survivorship analysis could not be performed; therefore, secondary efficacy/performance could not be assessed. It is to be noted that during the study, no intraoperative nor postoperative AEs were reported, as well as no reported subject deaths, therefore the raw survival for the 10 subjects in Arm B at the time of study closure was 100%.
Arm/Group | Arm B Reverse Shoulder Arthroplasty
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Collected from Baseline until study was terminated early (~24 Months).
Description: There were no Adverse Events Reported.
Arm/Group | Arm A Total Shoulder Arthroplasty / Hemiarthroplasty | Arm B Reverse Shoulder Arthroplasty
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/10
Other Adverse Events (participants affected / at risk) | 0/0 | 0/10

LIMITATIONS AND CAVEATS:
As the study was terminated early, outcomes and adverse events can only be reported up to the date of closure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT04089371/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-28): https://cdn.clinicaltrials.gov/large-docs/71/NCT04089371/SAP_001.pdf